CLINICAL TRIAL: NCT00966472
Title: A Phase I, Dose Finding Study of the Combination of High-dose Statin Agent (Rosuvastatin) With Erlotinib in Patients With Advanced Solid Malignancies, With a Focus on Squamous Cell Carcinomas and NSCLC.
Brief Title: Phase I Study of a Statin + Erlotinib for Advanced Solid Malignancies With Focus on Squamous Cell Carcinomas and NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007908-01H (OTT 08-07)
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Squamous Cell Carcinoma; Non-Small Cell Lung Cancer
Keywords: Rosuvastatin; Erlotinib; Squamous Cell Carcinoma; Nom-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib + Rosuvastatin (Experimental): To determine the recommended phase II dose (RP2D) of rosuvastatin that can be given in combination with standard erlotinib treatment in patients with advanced incurable squamous cell cancer and NSCLC.
  Interventions: Drug: Erlotinib + Rosuvastatin

INTERVENTIONS:
Drug: Erlotinib + Rosuvastatin — Patients will receive Erlotinib 150mg po daily. They will also receive Rosuvastatin at escalating dose levels starting at 1mg/kg po daily for 3 weeks, followed by a 1-week rest period. Patients may continue to receive rosuvastatin and erlotinib in the absence of disease progression or unacceptable toxicity.
  Other Names: Tarceva; Crestor

SUMMARY:
The purpose of this study is to determine the recommended phase II dose (RP2D) of rosuvastatin that can be given in combination with standard erlotinib treatment in patients with advanced incurable squamous cell cancer and NSCLC.

DETAILED DESCRIPTION:
Cytotoxic chemotherapy remains the mainstay of anti-cancer medical treatment for the vast majority of patients with locally advanced or metastatic squamous cell cancers. However, curative success remains low and most patients eventually succumb to the disease or its complications. Moreover, cytotoxic chemotherapy is frequently associated with severe unwanted side effects. Therefore, in this patient population the unmet therapeutic need is high and new treatment is required.

Statins are drugs which inhibit the cellular mevalonate pathway and are conventionally used in the treatment of hypercholesterolemia in cardiovascular disorders. Increasing evidence suggests that statins might be used for cancer prevention/treatment through their interactions with essential cellular functions, such as cell proliferation and differentiation. Recent in vitro data indicate that statins induce growth arrest and apoptosis, inhibit secretion of proteolytic enzymes, reduce invasiveness and inhibit angiogenesis. These effects contribute to the reduction of tumor growth and metastases in preclinical in vivo models of a variety of tumors suggesting that statins may be useful in anticancer therapy. Studies previously performed by our group demonstrated that targeting the mevalonate pathway can induce tumor specific cytotoxicity in a number of tumor types that included squamous cell carcinomas, myeloid leukemia and a variety of pediatric cancers. Additionally, several clinical trials have also assessed the antitumor activity of statins.

Pre-clinically, we have demonstrated additive cytotoxic effects when combining lovastatin with tyrosine kinase inhibitors of the Epidermal Growth Factor Receptor (EGFR) in HNSCC cells (AG1478) and in 8 squamous cell carcinomas (gefitinib). Mechanistically, lovastatin treatment inhibited EGF induced EGFR autophosphorylation by 24hrs and showed co-operative targeting of the EGFR in combination with gefitinib. Taken together, these results demonstrate that targeting the mevalonate pathway can inhibit EGFR function and suggest the potential utility of combining these classes of drugs (i.e. an EGFR tyrosine kinase inhibitor and a statin).

The use of lovastatin is not optimal due to greatly enhanced toxicity with drugs such as gefitinib and erlotinib that are simultaneously metabolized by the same enzyme (cytP450A4). In contrast, rosuvastatin a relatively novel potent mevalonate pathway inhibitor is not metabolized significantly by cytP450A4. Due to the enhanced clinical activity of erlotinib in comparison to other EGFR tyrosine kinase inhibitors, the combination of erlotinib and rosuvastatin appears ideal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented advanced and/or metastatic incurable tumor (especially squamous cell carcinoma or NSCLC).
* Clinically or radiologically documented (measurable or evaluable)disease.
* 18 years or older and less than 70 years of age.
* ECOG performance status: 0, 1 or 2
* No previous therapy with EGFR inhibitor (monoclonal antibody or TKI).
* Must have recovered from any treatment related toxicities prior to registration.
* Curative radiotherapy must be completed at least 3 months prior to registration
* Palliative radiotherapy is permitted providing a minimum of 14 days have elapsed between the end of radiotherapy and registration onto the study and patients have recovered from any acute toxic effects from radiation prior to registration.
* Previous surgery is permitted provided wound healing has occurred and at least 14 days have elapsed prior to registration if surgery was major.
* Adequate hematopoietic, hepatic and renal function defined as follows: hemoglobin >= 90g/L, platelets > 100 x 10^9/L, bilirubin <1.5 x ULN, ALT or AST <1.5 x ULN, proteinuria < grade 1, normal thyroid function (normal TSH or free T4 level after correction), serum creatinine institution normal limits or calculated creatinine clearance > 60 mls/min (except for patients with cervical cancer who require a creatinine clearance of 72 mls/min.)
* Women must be post menopausal, surgically sterile or use two reliable forms of contraception. Women of childbearing potential must have a serum or urine pregnancy test taken and proven negative within 7 days prior to registration. Men must be surgically sterile or use a barrier method of contraception
* Accessible for repeat dosing and follow-up

Exclusion Criteria:

* Asian ethnicity (Filipino, Chinese, Japanese, Korean, Vietnamese, or South Asian origin)
* History of other malignancies, except adequately treated non-melanoma skin cancer or other solid tumors curatively treated with no evidence of disease for > 5 years.
* Untreated brain or meningeal metastases. Patients with treated and radiologic or clinical evidence of stable brain metastases are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 4 weeks prior to registration).
* Untreated and/or uncontrolled cardiovascular conditions and/or symptomatic cardiac dysfunction.
* Active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Concurrent treatment with other experimental drugs or anti-cancer therapy.
* Patients who require oral anticoagulants (coumadin, warfarin) are eligible provided there is strict vigilance with respect to monitoring INR. The investigator should consider switching these patients to LMW heparin or an oral anti-platelet agent such as aspirin
* Patients who are taking concomitant medications, which are highly protein bound, nephrotoxic, or which are known strong inhibitors or inducers of the hepatic p450 (especially CYP3A4) system, which have not been discontinued prior to study registration. Caution should be exercised, and patients monitored closely, for patients taking concomitant drugs with the potential to inhibit or induce the hepatic p450 (especially CYP3A4) system.
* Any use of hypocholesterolemia agent such as niacin, fibrates or any statin should be discontinued at least 7 days prior to study registration.
* Personal or family history of hereditary muscular disorders
* Previous history of muscular toxicity with another HMG-CoA reductase inhibitor
* Alcohol abuse
* Any condition that could affect absorption of study oral drugs (erlotinib and rosuvastatin)
* Inflammatory bowel disease
* Uncontrolled hypothyroidism
* Chronic liver disease (ex: biliary sclerosis)
* Suffering from infection with HIV, Tuberculosis, Hepatitis C or Hepatitis
* Inability to give written, informed consent prior to study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the RPTD of rosuvastatin given orally daily x 3 weeks then 1 week off (28-day cycle) in combination with erlotinib given orally daily in patients with advanced solid tumors, especially squamous cell carcinomas and NSCLC. | Within 6 months
  To determine the RPTD of rosuvastatin

SECONDARY OUTCOMES:
To determine the safety, tolerability, toxicity profile, dose limiting toxicities and PK profile of rosuvastatin and erlotinib when given as combination therapy. | Within 6 months
  To determine the safety, tolerability, toxicity profile, dose limiting toxicities
To perform preliminary assessment of the anti-tumor activity of rosuvastatin in combination with erlotinib in patients with measurable disease. | Within one year
  To perform preliminary assessment of the anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Glenwood Goss, MD, FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Goss GD, Jonker DJ, Laurie SA, Weberpals JI, Oza AM, Spaans JN, la Porte C, Dimitroulakos J. A phase I study of high-dose rosuvastatin with standard dose erlotinib in patients with advanced solid malignancies. J Transl Med. 2016 Mar 31;14:83. doi: 10.1186/s12967-016-0836-6. PMID 27036206